CLINICAL TRIAL: NCT01245465
Title: Safety and Efficacy of Profermin® to Induce Remission in Patients With Ulcerative Colitis
Brief Title: Profermin® in Active Ulcerative Colitis
Acronym: CUPE-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nordisk Rebalance A/S (Industry)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Hans Israelsen, Noreba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-B-2008-FSP-20
Record Dates: First submitted 2010-11-18; First posted 2010-11-22 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — profermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Profermin (Experimental): Daily oral intake of a food for special medical purposes (Profermin)
  Interventions: Other: Profermin

INTERVENTIONS:
Other: Profermin — Medical Food (food for special medical purposes)

SUMMARY:
In this study the investigators aim was to investigate the safety and possible efficacy of Profermin® in patients with ulcerative colitis. The investigators also aimed at assessing the usefulness of a new online daily symptom registration system.

ELIGIBILITY:
Inclusion Criteria:Patients were eligible if they were between 18 and 50 years of age and had an established diagnosis of UC based on clinical, endoscopic and histological features. Active disease was assessed by Simple Clinical Colitis Activity Index (SCCAI) (Table 1) score above 4 and below 12.

-

Exclusion Criteria:

Patients who initiated treatment with azathioprine, 6-mercaptopurine, ciclosporin or methotrexate within 8 weeks prior to inclusion or TNF-α inhibitors within 12 weeks before inclusion or had changes in UC treatment within 2 weeks before inclusion were ineligible for the study. Concomitant coeliac disease or lactose intolerance were also exclusion criteria. In addition any malignant or premalignant condition or recent gastroenteritis rendered patients ineligible-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Our primary endpoint was to estimate the proportion of patients with a reduction in SCCAI ≥50%. | 24 weeks
  Daily report of SCCAI symptoms on the Internet

SECONDARY OUTCOMES:
Our secondary endpoint was to estimate the proportion of patients in remission defined as SCCAI lower than or equal to 2.5 | 24 weeks
  Daily report of SCCAI symptoms on the Internet

CONTACTS AND LOCATIONS:
Overall Officials: Hans Israelsen, PhD, Study Director — Nordisk Rebalance A/S